CLINICAL TRIAL: NCT03586843
Title: A Single-dose, Open-label, Randomized, 3-period, 6-sequence, Crossover Study to Evaluate the Relative Bioavailability of JNJ-64565111 After Single Subcutaneous Administration at Different Injection Sites in Otherwise Healthy Overweight/Obese Adult Subjects and A Multiple Dose, Open-label, Titration Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JNJ 64565111 in Otherwise Healthy Obese Adult Subjects
Brief Title: A Study of JNJ-64565111 After Single Subcutaneous Administration at Different Injection Sites in Otherwise Healthy Overweight/Obese Adult Participants and a Study of JNJ-6456511 in Otherwise Healthy Obese Adult Participants After Multiple Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108509; 64565111OBE1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-06-29; First posted 2018-07-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Treatment Sequence ABC: JNJ-64565111 (Experimental): Participants will receive Treatment A (JNJ-64565111 subcutaneous [SC] administration in the upper arm in fasted condition) on Day 1 of Treatment Period 1; followed by Treatment B (JNJ-64565111 SC administration in the thigh in fasted condition) on Day 1 of Treatment Period 2 and then Treatment C (JNJ-64565111 SC administration in the abdomen in fasted condition) on Day 1 of Treatment Period 3. Each treatment period will be separated by a washout Period of at least 7 days between the last pharmacokinetic (PK) sample collection and dosing on Day 1 of subsequent treatment period.
  Interventions: Drug: JNJ-64565111
- Part A: Treatment Sequence ACB: JNJ-64565111 (Experimental): Participants will receive Treatment A on Day 1 of Treatment Period 1; followed by Treatment C on Day 1 of Treatment Period 2 and then Treatment B on Day 1 of Treatment Period 3. Each treatment period will be separated by a washout Period of at least 7 days between the last PK sample collection and dosing on Day 1 of subsequent treatment period.
  Interventions: Drug: JNJ-64565111
- Part A: Treatment Sequence BAC: JNJ-64565111 (Experimental): Participants will receive Treatment B on Day 1 of Treatment Period 1; followed by Treatment A on Day 1 of Treatment Period 2 and then Treatment C on Day 1 of Treatment Period 3. Each treatment period will be separated by a washout Period of at least 7 days between the last PK sample collection and dosing on Day 1 of subsequent treatment period.
  Interventions: Drug: JNJ-64565111
- Part A: Treatment Sequence BCA: JNJ-64565111 (Experimental): Participants will receive Treatment B on Day 1 of Treatment Period 1; followed by Treatment C on Day 1 of Treatment Period 2 and then Treatment A on Day 1 of Treatment Period 3. Each treatment period will be separated by a washout Period of at least 7 days between the last PK sample collection and dosing on Day 1 of subsequent treatment period.
  Interventions: Drug: JNJ-64565111
- Part A: Treatment Sequence CAB: JNJ-64565111 (Experimental): Participants will receive Treatment C on Day 1 of Treatment Period 1; followed by Treatment A on Day 1 of Treatment Period 2 and then Treatment B on Day 1 of Treatment Period 3. Each treatment period will be separated by a washout Period of at least 7 days between the last PK sample collection and dosing on Day 1 of subsequent treatment period.
  Interventions: Drug: JNJ-64565111
- Part A: Treatment Sequence CBA: JNJ-64565111 (Experimental): Participants will receive Treatment C on Day 1 of Treatment Period 1; followed by Treatment B on Day 1 of Treatment Period 2 and then Treatment A on Day 1 of Treatment Period 3. Each treatment period will be separated by a washout Period of at least 7 days between the last PK sample collection and dosing on Day 1 of subsequent treatment period.
  Interventions: Drug: JNJ-64565111
- Part B: JNJ-64565111 (Experimental): Participants will receive a single SC ascending doses of JNJ-64565111 on Days 1, 8, 15, 22, 29 and 36.
  Interventions: Drug: JNJ-64565111

INTERVENTIONS:
Drug: JNJ-64565111 — JNJ-64565111 SC will be administered on Day 1 of Treatment Periods 1, 2 and 3 as per the assigned treatment sequence in Part A and as ascending doses on Days 1, 8, 15, 22, 29 and 36 in Part B.

SUMMARY:
The purpose of this study is to compare the relative bioavailability of JNJ-64565111 between subcutaneous (SC) administrations in the upper arm versus the abdomen, and between SC administrations in the thigh versus the abdomen in otherwise healthy overweight/obese participants (Part A) and to assess the gastrointestinal tolerability of JNJ-64565111 following a dose titration in otherwise healthy obese participants at 6 weeks (Part B).

ELIGIBILITY:
Inclusion Criteria:

Part A and Part B:

- If a woman, must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry, throughout the study and for at least 30 days after the last dose of study drug

Part A:

* If a woman, must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test at screening; and a negative serum pregnancy test on Day -1 of each treatment period
* Body mass index (weight [kilogram {kg}]/height^2 [meter {m}^2]) between 25-40 kg/m^2 (inclusive), and body weight not less than 75 kg

Part B:

* A woman must have a negative serum beta-hCG pregnancy test at screening, on Day 1, and before each SC injection, except on Day 8(+1). On Day 8(+1), women must have a negative serum or urine pregnancy test depending on the test performed at the investigator's discretion
* Body mass index (weight [kg]/height^2 [m]^2) between 30-50 kg/m^2 (inclusive), and body weight not less than 75 kg

Exclusion Criteria:

Part A and Part B:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities (that is [ie], fasting triglycerides greater than or equal to (>=)500 milligram per deciliter (mg/dL) and/or total cholesterol >=300 mg/dL), significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at screening or at admission to the study center as deemed appropriate by the investigator
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study center as deemed appropriate by the investigator. Participants with serum sodium less than (<)130 milliequivalents per liter (mEq/L) at screening should be excluded
* Known allergy to the study drug or any of the excipients of the formulation
* Donated blood or blood products or had substantial loss of blood (more than 500 milliliters [mL]) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study or within 2 months after the completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Serum Concentration of JNJ-64565111 (Cmax) | Predose, 4, 8, 12, 24, 36, 48, 72, 96, 144, 192, 384, 672 and 984 hours postdose; at End of study (EOS): 7-14 days after Day 42 of Treatment Period 3 (approximately up to 26 weeks)
  Cmax is the maximum observed serum analyte concentration.
Part A: Area Under the Serum Concentration Time Curve From Time 0 to Infinite Time (AUC [0-infinity]) | Predose, 4, 8, 12, 24, 36, 48, 72, 96, 144, 192, 384, 672 and 984 hours postdose; at EOS: 7-14 days after Day 42 of Treatment Period 3 (approximately up to 26 weeks)
  AUC [0-infinity) is the area under the serum concentration versus time curve from time 0 to infinite time, calculated as AUClast + Clast/lambda(z) where Clast is the last observed measurable (non- below quantification limit [BQL]) concentration.
Part A: Area Under the Serum Concentration Time Curve From Time 0 to Time of the Last Measurable Concentration (AUC [0-last]) | Predose, 4, 8, 12, 24, 36, 48, 72, 96, 144, 192, 384, 672 and 984 hours postdose; at EOS: 7-14 days after Day 42 of Treatment Period 3 (approximately up to 26 weeks)
  AUC (0-last) is the area under the serum concentration versus time curve from time 0 to time of the last measurable (non-below quantification limit [BQL]) concentration, calculated by linear linear trapezoidal summation.
Part B: Number of Participants with Gastrointestinal Adverse Events as a Measure of Safety and Tolerability of JNJ-64565111 | Approximately up to 6 weeks
  Number of participants with gastrointestinal adverse events will be assessed. An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily have a causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Part A and Part B: Number of Participants with Antibodies to JNJ-64565111 | Part A: Predose, 144, 672 and 984 hours postdose; at EOS: 7-14 days after Day 42 of Treatment Period 3 (approximately up to 26 weeks); Part B: predose (Day 1), postdose on Day 39 or End of Study/Early Withdrawal (approximately up to 7 weeks)
  Number of participants with antibodies to JNJ-64565111 will be reported.
Part A and Part B: Number of Participants with Adverse Events | Part A: approximately up to 26 weeks, Part B: approximately up to 11 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily have a causal relationship with the relevant investigational product.
Part B: Number of Gastrointestinal Adverse Events Over Time Upon Multiple Dosing | Approximately up to 6 weeks
  The number of gastrointestinal adverse events over time will be evaluated upon multiple dosing of JNJ-64565111.
Part B: Maximum Observed Serum Concentration of JNJ-64565111 (Cmax) | From Day 36 until Day 43
  Cmax (maximum observed serum analyte concentration) after last dose of JNJ-64565111.
Part B: Area Under the Serum Concentration Versus Time Curve Over the Dosing Interval (AUCtau) | From Day 36 until Day 43
  AUCtau (measure of the serum drug exposure over the dosing interval) after the last dose of JNJ-64565111.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Celerion, Tempe, Arizona, United States